CLINICAL TRIAL: NCT07035210
Title: Impact of Self-directed Goals for Long-term Patients in a Forensic Hospital: A Mixed-Methods Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chapin Graham (Other)
Responsible Party: Sponsor-Investigator, Chapin Graham, Occupational Therapy Doctoral Student, Johnson & Wales University
Organization: Johnson & Wales University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPA#241002
Record Dates: First submitted 2025-02-27; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-02

CONDITIONS: Occupational Deprivation; Forensic Mental Health
Keywords: Long-term patients; Forensic patients; Mental health patients; Occupational deprivation; Self-directed goals
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-directed Goals (Experimental): Participants will be setting self-directed goals based on the Canadian Occupational Performance Measure in skilled 1:1 occupational therapy sessions and working to achieving them as well as attending a goal-setting educational group.
  Interventions: Behavioral: Group and 1:1 occupational therapy sessions

INTERVENTIONS:
Behavioral: Group and 1:1 occupational therapy sessions — Patients will be educated on the goal setting process and setting self-directed goals aimed at occupations they identified as important in both group and 1:1 treatment sessions.

SUMMARY:
The goal of this study is to determine if supporting forensic patients in setting their own goals can impact occupational deprivation. This study is guided by this overarching research question: can setting and achieving self-directed goals improve occupational deprivation outcomes in long-term patients of a forensic psychiatric hospital? Participants were provided an educational group and occupational therapy treatment sessions to support goal setting within the forensic hospital.

DETAILED DESCRIPTION:
The forensic hospital in which this research will be completed has patients with one of the following statuses:

* Incompetent to stand trial (IST): these patients are pretrial detainees with criminal charges who come from the department of corrections (DOC) remanded by the courts for psychiatric treatment and competency to stand trial restoration. Incompetent to stand trial means a patient is unable to participate in the court proceedings due to active symptoms of mental illness. Once recommended as competent, they can move forward to face their charges and hopefully be discharged from the hospital.
* Specialized services (SS): Patients admitted on SS are serving a sentence. While they are at the DOC, symptoms of their mental illness either emerge or get worse, impacting their safety to the extent that they need a hospital level of psychiatric care that cannot be provided in a correctional setting.
* Not guilty by reason of insanity (NGRI): A patient who has gone through the court process and adjudicated as NGRI. They have been committed to the department of mental health and reside in a forensic hospital. While there, they will continue to receive treatment and achieve incremental privileges approved first by the Psychiatric Services Review Board (PSRB) then by the court. They remain at the forensic hospital to serve time until they are up for parole.

The participants in the study will have a variety of these statuses. The population of long-term patient participants for this study are defined as having been hospitalized for at least one year at the start date of recruitment with no imminent discharge date. The participants will be assessed by the Canadian Occupational Performance Measure (COPM) before the first week of treatment to determine occupations they want to set goals for, and determine how they are currently performing those occupations as well as how satisfied they are with that performance. The project site has the COPM, so there is no funding necessary. The COPM can also be administered by any occupational therapist familiar with the assessment, so no additional training is necessary. After 10 weeks of treatment, the COPM will be used as a post-test as well.

Treatment includes: ten 1:1 occupational therapy sessions to achieve these goals and a ten week group with the focus of education on the goal-setting process. It is hypothesized that they will see improvement in satisfaction of the occupations they set goals around. It should be noted that all participants will have treatment goals set by the occupational therapy (OT) department that will be tracked and documented in the patients' medical chart, as is routine for OT treatment and per OT department policy.

Patient scores of performance and satisfaction will be compared between the first and second trial. Score changes are clinically significant if it is a change of two points or higher. To support the findings, patients' self-directed goals, when they are achieved, and any statements related to the setting and achieving of goals will be collected for qualitative analysis. This analysis and data will be deidentified using participant numbers and stored on a password protected Google Drive that can only be accessed by investigator (Chapin Graham) and site mentor (Natalie Petrucci). Hard copies of the COPM will be shredded once scanned into the Google Drive. All information on the Google Drive will be moved to trash and then the trash folder will be cleared one year after completion of the study.

Patients have the ability to leave the study at any time with no negative repercussions by simply refusing 1:1 treatment or group sessions. If they decompensate and exhibit psychotic behaviors, they will be discharged from the study involuntarily with no negative repercussions. Since the patients are their own legal guardians, they are fit to make informed consent for treatment at the hospital, including participation in this study.

Participant expectations

Participants will engage in assessment, evaluation, and treatment. The assessment and evaluations will serve to tailor their treatment to their current level of need. They will work with the OTS to schedule a weekly meeting time and, if a part of the variable group, attend all 10 weeks of the group. These sessions can be flexible based on hospital events, unexpected visits, or other conflicts. The expectations of the control group will be the same as the variable group, except for the attendance of the goal education group.

Data Collection

Assessment and evaluation will consist of the COPM and an in depth chart review to determine current level of function. The assessment write up, goals, 1:1 treatment notes and group notes will become part of the patient's medical record that is saved on the hospital encrypted drive. There will also be data that is collected solely for the purpose of the research, such as COPM scores, self-directed goals set, when the goals are achieved, and any quotes surrounding the goal-setting process.

This data will be stripped of identifying information and stored on a password protected Google Drive. Clients will be assigned a number and referred only by this. There will be no information related to birthday, age, hospital status, diagnosis, or criminal case. The only people with access will be the investigator (Chapin Graham) and site mentor (Natalie Petrucci). One year after the completion of the study, records on Google Drive will be moved to the trash folder and the trash folder will then be cleared, effectively destroying the records.

In order to be included in the study, patients will provide informed consent and be made aware that they are able to terminate their participation without any repercussions to their current treatment.

The routine of the hospital allows for participation in referral-based groups and patient treatment on occupational therapy caseload, assuring confidential participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Is capable of providing consent to participate.
* Is at least 18 years of age.
* Resides at Rhode Island State Psychiatric Hospital.
* Hospital stay for a year or longer as of the anticipated start date of January 2025.
* No imminent discharge date due to the nature of their alleged criminal charges or current symptoms of their mental illness.

Exclusion Criteria:

* Have an imminent discharge date
* Having experienced positive symptoms of psychosis (i.e hallucinations, delusions, or thought disorganization) in the year prior to the January start date.
* Behavioral outburst resulting in restraints in the year prior to the January start date.
* Hold a primary diagnosis of antisocial personality disorder (ASPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | At enrollment and week 11
  Semi-structured interview identifying occupational participation. Participants rate occupations identified based on importance, performance, and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island State Psychiatric Hospital, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephenson T, Leaman J, O'Moore E, Tran A, Plugge E. Time out of cell and time in purposeful activity and adverse mental health outcomes amongst people in prison: a literature review. Int J Prison Health. 2021 Jan 6;17(1):54-68. doi: 10.1108/IJPH-06-2020-0037. PMID 33634654
- [Background] Romero-Ayuso DM, Toledano-Gonzalez A, Pinilla-Cerezo M, Sanchez-Rodriguez O, Garcia-Arenas JJ, Trivino-Juarez JM, Ortiz-Rubio A. Occupational Balance and Emotional Regulation in People With and Without Serious Mental Illness. Can J Occup Ther. 2024 Mar;91(1):100-109. doi: 10.1177/00084174231178440. Epub 2023 Jun 4. PMID 37271981
- [Background] Law M, Polatajko H, Pollock N, McColl MA, Carswell A, Baptiste S. Pilot testing of the Canadian Occupational Performance Measure: clinical and measurement issues. Can J Occup Ther. 1994 Oct;61(4):191-7. doi: 10.1177/000841749406100403. PMID 10137673
- [Background] Laverdure P, Beisbier S. Occupation- and Activity-Based Interventions to Improve Performance of Activities of Daily Living, Play, and Leisure for Children and Youth Ages 5 to 21: A Systematic Review. Am J Occup Ther. 2021 Jan-Feb;75(1):7501205050p1-7501205050p24. doi: 10.5014/ajot.2021.039560. PMID 33399053
- [Background] Clarke, C. (2003). Clinical application of the Canadian Model of Occupational Performance in a forensic rehabilitation hostel. British Journal of Occupational Therapy, 66(4).